CLINICAL TRIAL: NCT04552847
Title: Al18F-NOTA-octreotide PET Imaging of the Somatostatin Receptor in Neuroendocrine Tumors
Brief Title: Al18F-NOTA-octreotide PET Imaging in Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Hospital, Antwerp (Other); University Hospital, Ghent (Other); NETwerk, Belgium (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S63678
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Neuroendocrine Tumors
Keywords: Somatostatin receptor imaging; Al18F-NOTA-octreotide; PET/CT; PET/MR
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Al18F-NOTA-octreotide; Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): In the main part of the trial (part A) 75 patients with cytologically and/or histologically confirmed neuroendocrine tumors of all grades of gastroenteropancreatic, pulmonary, neural crest or unknown primary origin will receive a single intravenous injection of Al18F-NOTA-octreotide. At two hours after tracer injection they will undergo a whole-body PET/CT scan.
  In part B of the trial 10 up to 20 patients with with cytologically and/or histologically confirmed neuroendocrine tumors of all grades of gastroenteropancreatic, pulmonary, neural crest or unknown primary origin will receive a single intravenous injection of Al18F-NOTA-octreotide. At two hours after tracer injection they will undergo a whole-body PET/MR scan.
  Interventions: Drug: Al18F-NOTA-octreotide; Device: PET/CT; Device: PET/MR

INTERVENTIONS:
Drug: Al18F-NOTA-octreotide — One intravenous injection of 4 MBq/kg
  Other Names: 18F-AlF-NOTA-octreotide; 18F-IMP-466
Device: PET/CT — Patients in part A of the trial will undergo a whole-body PET/CT scan 120 minutes (acceptable range: 105 - 240 minutes) after injection of the tracer. The CT-scan is a low-dose CT that will be acquired for both PET attenuation correction and anatomical information.
Device: PET/MR — Patients in part B of the trial will undergo a whole-body PET/MR scan 120 minutes (acceptable range: 105 - 240 minutes) after injection of the tracer. The MR scan is a fully diagnostic MR requiring intravenous contrast (Dotarem®) injection and Buscopan® administration to minimize bowel movement.

SUMMARY:
The aim of this study is to evaluate the diagnostic performance of Al18F-NOTA-octreotide PET imaging in comparison with the current golden standard, 68Ga-DOTA-somatostatin analog PET, in neuroendocrine tumor patients.

DETAILED DESCRIPTION:
Part A (main part of the trial):

Seventy-five neuroendocrine tumor (NET) patients (M/F, aged 18 years and older) with a routine clinical 68Ga-DOTA-somatostin analog (SSA) PET/CT performed in the last three months or scheduled within three months, will undergo a whole-body Al18F-NOTA-octreotide PET/CT.

Part B:

At least 10, possibly up to 20 NET patients (M/F, aged 18 years and older) with a routine clinical 68Ga-DOTA-SSA PET/CT performed in the last three months or scheduled within three months, will undergo a whole-body Al18F-NOTA-octreotide PET/MR.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged over 18 years.
* Signed Informed Consent.
* Subject is diagnosed with a histologically and/or cytologically confirmed neuroendocrine tumor of all grades of gastroenteropancreatic, pulmonary, neural crest or unknown primary origin.
* Subject should have at least one known tumoral lesion below the level of the submandibular and parotid glands with either a minimum size of 1 cm in at least one dimension on morphological imaging (CT, MRI, ultrasound), or a maximal standardized uptake value (SUVmax) of at least 10 on 68Ga-DOTA-SSA PET, in both cases performed within 4 months prior to study scan. A positive lesion is defined as a volume of increased tracer uptake compared to background, deemed to be caused by the presence of NET cells, and that is unlikely to be attributed to physiological or benign etiology (e.g. inflammation, blood pool retention, excretion, etc.).
* Subject should have a routine clinical 68Ga-DOTA-SSA PET/CT performed within three months prior to the study scan or scheduled within three months after the study scan.
* Female subjects should be (a) post-menopausal, or (b) surgically sterile, or (c) using effective contraceptive with negative pregnancy test.

Exclusion Criteria:

Part A and B:

* Subject has a previous or ongoing recurrent or chronic disease, other than a neuroendocrine tumor, at high risk to interfere with the performance or evaluation of the trial according to the judgement of the investigator.
* Subject has had exposure to ionizing radiation (> 1 mSv) in other research studies within the last 12 months.
* Subject has recently (< 30 days or 5 times the plasma half-life of the investigated drug, whichever is longest) participated or is simultaneously participating in another prospective interventional clinical trial.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e. weight lifting, running, bicycling) beginning 4 days prior to tracer injection up to 1 day after tracer injection.
* Subject is potentially pregnant (urinary hCG test can be performed in case of doubt) or is breast-feeding.
* Subject is unwilling or unable to perform all of the study procedures, or is considered unsuitable in any way by the principal investigator.
* Subject does not understand the study procedure.
* Subject is mentally or legally incapacitated.

Only for part B:

* Subject has a contra-indication for MR scanning.
* Subject suffers from claustrophobia or cannot tolerate confinement during PET/MR scanning.
* Subject has an impaired renal function: estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m² (the last known value may not date from more than 3 months prior to the study PET/MR; if not available a blood analysis may be performed as part of the trial).
* Subject suffers from diseases for which butylhyoscine bromide (Buscopan®) is contra-indicated: glaucoma, paralytic ileus, severe colitis ulcerosa or myasthenia gravis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Differential detection ratio (DDR) | 2 years
  The fraction of lesions detected by one tracer is the detection ratio. In case of non-inferiority, the difference in detection ratio on Al18F-NOTA-octerotide PET and the detection ratio on 68Ga-DOTA-SSA PET, i.e. the differential detection ratio (DDR), equals zero. The primary objective will be met if the lower margin of the 95% confidence interval for the DDR is higher than -15%. Readers will be blinded for the radiopharmaceutical that is used. (only for part A of the trial)

SECONDARY OUTCOMES:
Lesion detection rate on the organ level | 2 years
  A sub analysis will be performed, involving a lesion count per organ to determine the sensitivity of Al18F-NOTA-octreotide PET and 68Ga-DOTA-SSA PET on the organ level.
Lesion uptake | 2 years
  Standardized uptake value (SUV) measurements will be performed: SUVmax for lesions and SUVmean for several background areas will be determined. Lesion uptake, in terms of SUVmax and tumor-to-background ratio (TBR), will be compared for both tracers.
Clinical impact on TNM staging or patient management | 2.5 years
  We will evaluate whether different findings with both tracers have a clinical impact, e.g. leading to different TNM staging or differences in patient management. (only part A of the trial as this will be blinded)
Lesion detection rate according to the specific 68Ga-DOTA-SSA used for the routine PET scan | 2 years
  Due to the multicenter nature of this study, two or three different standard PET tracers will be used for the routine clinical care 68Ga-DOTA-SSA PET: 68Ga-DOTATATE (current standard in UZ Leuven), 68Ga-DOTANOC (current standard in UZ Antwerp), and potentially 68Ga-DOTATOC (depending where patients from UZ Ghent are scanned). Therefore, the diagnostic performance of Al18F-NOTA-octreotide PET will also be compared with the two or three 68Ga-DOTA-SSAs tracers separately.
Lesion detection rate according to tumor grade | 2 years
  A sub analysis will be performed, comparing the diagnostic performance and lesion uptake with Al18F-NOTA-octreotide and 68Ga-DOTA-SSA between low-grade and high-grade NETs.
Overall diagnostic image quality according to a five-point Likert-scale | 3 years
  As part of an inter-observer agreement analysis, readers will score overall diagnostic image quality using a five-point Likert-scale: (1) non diagnostic, (2) poor, (3) sufficient, (4) good and (5) excellent.
Lesion conspicuity according to a five-point Likert-scale | 3 years
  As part of an inter-observer agreement analysis, readers will score lesion conspicuity relative to the surrounding background using a five-point Likert-scale: (1) no increased uptake (equal or lower than background uptake), (2) barely perceived (slightly higher than background uptake), (3) moderately detectable (higher than background uptake, but less than twice, or less than 5 standardized uptake value (SUV) units above, the background uptake), (4) definitely detected (at least twice the background uptake and at least 5 SUV units higher than background uptake) and (5) strikingly evident/easily spotted (evident on maximum intensity projection images and typically higher than uptake in all normal organs, including the spleen).
Diagnostic confidence according to a five-point Likert-scale | 3 years
  As part of an inter-observer agreement analysis, for each focus of increased non-physiologic uptake readers will score diagnostic confidence using a five-point Likert-scale: (1) definitely no lesion, (2) probably no lesion, (3) indeterminate, (4) probably a lesion, (5) definitely a lesion.
Whole-body MRI correlate of the lesions detected by the PET scans | 2.5 years
  For the union of lesions identified on both PET scans, MRI images will be checked for corresponding MRI lesions. If a correlating lesion is detected and deemed to be of malignant nature by an experienced whole-body MRI radiologist, the PET lesions will be considered true positives. (only part B of the trial)
Effect of Al18F-NOTA-octreotide injection on blood pressure | 2 years
  The impact of Al18F-NOTA-octreotide administration on blood pressure (in mmHg) will be assessed. This parameter and changes from baseline values will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Effect of Al18F-NOTA-octreotide injection on heart rate | 2 years
  The impact of Al18F-NOTA-octreotide administration on heart rate (in beats per minute) will be assessed. This parameter and changes from baseline values will be scored according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Deroose, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pauwels E, Cleeren F, Tshibangu T, Koole M, Serdons K, Dekervel J, Van Cutsem E, Verslype C, Van Laere K, Bormans G, Deroose CM. [18F]AlF-NOTA-octreotide PET imaging: biodistribution, dosimetry and first comparison with [68Ga]Ga-DOTATATE in neuroendocrine tumour patients. Eur J Nucl Med Mol Imaging. 2020 Dec;47(13):3033-3046. doi: 10.1007/s00259-020-04918-4. Epub 2020 Jul 2. PMID 32617641
- [Derived] Leupe H, Pauwels E, Vandamme T, Van den Broeck B, Lybaert W, Dekervel J, Van Herpe F, Jaekers J, Cleeren F, Hofland J, Brouwers A, Koole M, Bormans G, Van Cutsem E, Geboes K, Laenen A, Verslype C, Stroobants S, Deroose CM. Clinical impact of using [18F]AlF-NOTA-octreotide PET/CT instead of [68Ga]Ga-DOTA-SSA PET/CT: Secondary endpoint analysis of a multicenter, prospective trial. J Neuroendocrinol. 2024 Aug;36(8):e13420. doi: 10.1111/jne.13420. Epub 2024 Jun 4. PMID 38837825
- [Derived] Boeckxstaens L, Pauwels E, Vandecaveye V, Deckers W, Cleeren F, Dekervel J, Vandamme T, Serdons K, Koole M, Bormans G, Laenen A, Clement PM, Geboes K, Van Cutsem E, Nackaerts K, Stroobants S, Verslype C, Van Laere K, Deroose CM. Prospective comparison of [18F]AlF-NOTA-octreotide PET/MRI to [68Ga]Ga-DOTATATE PET/CT in neuroendocrine tumor patients. EJNMMI Res. 2023 Jun 1;13(1):53. doi: 10.1186/s13550-023-01003-3. PMID 37261615
- [Derived] Pauwels E, Cleeren F, Tshibangu T, Koole M, Serdons K, Boeckxstaens L, Dekervel J, Vandamme T, Lybaert W, den Broeck BV, Laenen A, Clement PM, Geboes K, Cutsem EV, Stroobants S, Verslype C, Bormans G, Deroose CM. 18F-AlF-NOTA-Octreotide Outperforms 68Ga-DOTATATE/NOC PET in Neuroendocrine Tumor Patients: Results from a Prospective, Multicenter Study. J Nucl Med. 2023 Apr;64(4):632-638. doi: 10.2967/jnumed.122.264563. Epub 2022 Oct 20. PMID 36265911